CLINICAL TRIAL: NCT06051435
Title: Effect of Lumbar Proprioception Training on Primary Dysmenorrhea: A Randomized Clinical Trial
Brief Title: Effect of Lumbar Proprioception Training on Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa A. Osman, Assistant professor Physical Therapy for Woman's Health Faculty of Physical Therapy Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004410
Record Dates: First submitted 2023-09-11; First posted 2023-09-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Primary Dysmenorrhea
Keywords: lumbar proprioception training; pelvic rocking exercises; primary dysmenorrhea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): They will receive hot packs and pelvic rocking exercises for one menstrual cycle.
  Interventions: Other: Hot packs; Other: Pelvic rocking exercise
- Lumbar proprioception group (Experimental): They will receive the same lumbar proprioception training plus hot packs and pelvic rocking exercises for one menstrual cycle.
  Interventions: Other: lumbar proprioception training; Other: Hot packs; Other: Pelvic rocking exercise

INTERVENTIONS:
Other: lumbar proprioception training — a) Sensorimotor training: Sensorimotor training and reconditioning of proprioceptive senses have recently been found to be helpful in increasing motor performance and coordination, muscle strength, sensorimotor abilities, increasing intermuscular control, and improving one's response to sensory information and muscle tone. Reconditioning of proprioceptive senses and sensorimotor training increases one's muscle adjustment ability, maximizes the sensory input in different parts of the body and aids in improving one's motor adjustment ability (Hwang et al ., 2013).
  Position Exercise methods as Hollowing exercise: Participants will be asked to contract the abdominal muscles, raising the center of movement toward the navel in a quadruped position.
  Other Names: lumbar proprioception exercises
  Arms: Lumbar proprioception group
Other: Hot packs — hot application in the form of hot packs on the lower abdomen and lower back for a total duration of 30 minutes, once per day, during the first two days of menstruation
Other: Pelvic rocking exercise — Pelvic rocking exercise

SUMMARY:
the aim of this study will be to investigate the effect of lumbar proprioception training on primary dysmenorrhea.

DETAILED DESCRIPTION:
Although previous studies reported the effect of physiotherapy practices through therapeutic exercises on primary dysmenorrhea as core muscles strengthening, core stability exercises, connective tissue massage and classical massage, relaxation, strengthening, stretching, aerobic exercises, pelvic floor muscle strengthening exercises, yoga and Pilates. None of them have investigated the effect of lumbar proprioception training on primary dysmenorrhea. Therefore, this study will be the first one which aims to investigate the effect of lumbar proprioception training on primary dysmenorrhea. This trial will include 2 groups; group A composed of 20 females that will receive hot packs and pelvic rocking exercises for 4 weeks and group B also composed of 20 females that will receive hot packs and pelvic rocking exercises in addition to lumbar proprioception training for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All females will have moderate to severe primary dysmenorrhea (as determined by WaLIDD Scale).
* Their ages will range from 18 to 22 years old.
* All females will be virginal and non-smokers.
* Their BMI will be range from 20-25 kg/m2
* They have regular menstrual cycle with menstrual cycle length of 28-30 days.
* They have persistent primary dysmenorrhea of more than 6 months

Exclusion Criteria:

* They shouldn't have musculoskeletal or neurological disorders, chronic LBP or sacroiliac dysfunction, diabetes, pelvic pathology or any gynecological disease.
* They shouldn't experience a stressful event in the last 6 month.
* Attending regular exercise training in the last 6 months.
* Taking medications or vitamin and mineral supplements due to other medical conditions.

Ages: 18 Years to 22 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Measurement of lumbar proprioception | 4 weeks
  It will be evaluated through Biodex system in both groups before and after treatment program through measuring the lumbar repositioning accuracy.

SECONDARY OUTCOMES:
Calculation of score of WaLIDD Scale | 4 weeks
  It will be used to identify dysmenorrhea severity in both groups before and after treatment program through measuring combination of manifestations: subjective (intensity/Wong-Baker, work ability) and objective (days of pain, location) for both groups.The total score of 0 indicates without dysmenorrhea; 1-4 indicates mild dysmenorrhea, 5-7 indicates moderate dysmenorrhea, 8-12 indicates severe dysmenorrhea (Teherán et al., 2018).
lumbar curvature angle | 4 weeks
  it will be measured by Flexible ruler which is affected by the tilt of the pelvis, in both groups before and after treatment program.

CONTACTS AND LOCATIONS:
Overall Officials: Amel Mohamed Yousef, PhD, Study Chair — Professor, Cairo university; Hamada Ahmed Hamada, PhD, Study Director — Assistant Professor, Cairo university
Locations (1):
- Doaa Osman, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No